CLINICAL TRIAL: NCT04756050
Title: Comparison of Different Approaches for Supraclavicular Block and Their Effects on Diaphragm Muscle Function Evaluated With Diaphragm Thickening Fraction
Brief Title: Comparison of Different Approaches for Supraclavicular Block and Their Effects on Diaphragm Muscle Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Çağrı Yeşilnacar, anesthesiology resident, Bozyaka Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: cagritez
Record Dates: First submitted 2021-02-08; First posted 2021-02-16 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Phrenic Nerve Paralysis; Diaphragm Sellae Meningioma; Complications; Respiratory Complication; Nerve Block; Brachial Plexus Block
Keywords: Brachial Plexus Block; Phrenic Nerve Paralysis; Respiratory Complication; Complications; nerve block; Diaphragm
MeSH Terms: interventions — Bupivacaine; High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Three groups involved. 3 different approaches of supraclavicular block will be compared. Approaches share the same probe position and needle entry point but differ in where the local anesthetic is given.
  Group 1: Local anesthetic mixture will be given to the corner pocket - where the artery and the first rib intersect in the sonoanatomical image.
  Group 2: 10 ml of the local anesthetic mixture will be given to the described corner pack and the remaining 10 ml into the largest nerve cluster (Intracluster injection).
  Group 3: Local anesthetic mixture will be administered by multi injection method between the nerve groups seen in the sonoanatomical image.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant will not know which group he or she is in. The diaphragm thickening fraction and evaluations (outcomes) will be made by another experienced anesthesiologist, double-blindness will be achieved by being blind to the patient's group.
  Block evaluation and measurements will be made by a different experienced anesthesiologist .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- corner pocket (Experimental): The block will be performed by an experienced anesthesiologist in block applications under USG guidance. After the antisepsis of the area to be blocked, a 22G 50 mm stimulator needle will be used for the block . Intermittent negative aspiration will be performed during all procedures to detect possible vascular puncture. 20 ml of bupivacaine(Buvicaine HCl %0.5) and prilocaine(Priloc HCl %2) 1:1 mixture will be prepared in a way that there will be 5mcg adrenaline per ml.(9ml bupivacaine, 9ml prilocaine and 2ml saline with 50 mcg adrenaline per ml) Local anesthetic mixture will be given to the corner pocket - where the artery and the first rib intersect in the sonoanatomical image.
  Interventions: Drug: Bupivacaine HCl 0.5% Injectable Solution; Drug: Prilocaine HCl % 2 injectable solution; Drug: adrenaline amp 0.5mg; Procedure: Ultrasound Guided Supraclavicular Block Corner pocket approach; Procedure: diagraphma muscle evaluation with ultrasound
- corner+intracluster (Experimental): The block will be performed by an experienced anesthesiologist in block applications under USG guidance. After the antisepsis of the area to be blocked, a 22G 50 mm stimulator needle will be used for the block . Intermittent negative aspiration will be performed during all procedures to detect possible vascular puncture20 ml of bupivacaine(Buvicaine HCl %0.5) and prilocaine(Priloc HCl %2) 1:1 mixture will be prepared in a way that there will be 5mcg adrenaline per ml.(9ml bupivacaine, 9ml prilocaine and 2ml saline with 50 mcg adrenaline per ml) 10 ml of the local anesthetic mixture will be given to the described corner pack and the remaining 10 ml into the largest nerve cluster (Intracluster injection).
  Interventions: Drug: Bupivacaine HCl 0.5% Injectable Solution; Drug: Prilocaine HCl % 2 injectable solution; Drug: adrenaline amp 0.5mg; Procedure: Ultrasound Guided Supraclavicular Block Corner pocket + intracluster approach; Procedure: diagraphma muscle evaluation with ultrasound
- multi (Experimental): The block will be performed by an experienced anesthesiologist in block applications under USG guidance. After the antisepsis of the area to be blocked, a 22G 50 mm stimulator needle will be used for the block . Intermittent negative aspiration will be performed during all procedures to detect possible vascular puncture. 20 ml of bupivacaine(Buvicaine HCl %0.5) and prilocaine(Priloc HCl %2) 1:1 mixture will be prepared in a way that there will be 5mcg adrenaline per ml.(9ml bupivacaine, 9ml prilocaine and 2ml saline with 50 mcg adrenaline per ml) Local anesthetic mixture will be administered by multi injection method between the nerve groups seen in the sonoanatomical image.
  Interventions: Drug: Bupivacaine HCl 0.5% Injectable Solution; Drug: Prilocaine HCl % 2 injectable solution; Drug: adrenaline amp 0.5mg; Procedure: Ultrasound Guided Supraclavicular Block multi approach; Procedure: diagraphma muscle evaluation with ultrasound

INTERVENTIONS:
Drug: Bupivacaine HCl 0.5% Injectable Solution — 20 ml of bupivacaine(Buvicaine HCl %0.5) and prilocaine(Priloc HCl %2) 1:1 mixture will be prepared in a way that there will be 5mcg adrenaline per ml.(9ml bupivacaine, 9ml prilocaine and 2ml saline with 50 mcg adrenaline per ml)
  Other Names: buvicaine %0.5,
Drug: Prilocaine HCl % 2 injectable solution — 20 ml of bupivacaine(Buvicaine HCl %0.5) and prilocaine(Priloc HCl %2) 1:1 mixture will be prepared in a way that there will be 5mcg adrenaline per ml.(9ml bupivacaine, 9ml prilocaine and 2ml saline with 50 mcg adrenaline per ml)
  Other Names: priloc %2
Drug: adrenaline amp 0.5mg — 20 ml of bupivacaine(Buvicaine HCl %0.5) and prilocaine(Priloc HCl %2) 1:1 mixture will be prepared in a way that there will be 5mcg adrenaline per ml.(9ml bupivacaine, 9ml prilocaine and 2ml saline with 50 mcg adrenaline per ml)
  Other Names: adrenalin codex 0.5mg/1ml injectable solution
Procedure: Ultrasound Guided Supraclavicular Block Corner pocket approach — The blocks will be performed by an experienced anesthesiologist with a USG guidance. Local anesthetic mixture will be given to the corner pocket - where the artery and the first rib intersect in the sonoanatomical image.
  Arms: corner pocket
Procedure: Ultrasound Guided Supraclavicular Block Corner pocket + intracluster approach — The blocks will be performed by an experienced anesthesiologist with a USG guidance .10 ml of the local anesthetic mixture will be given to the described corner pack and the remaining 10 ml into the largest nerve cluster (Intracluster injection).
  Arms: corner+intracluster
Procedure: Ultrasound Guided Supraclavicular Block multi approach — The blocks will be performed by an experienced anesthesiologist with a USG guidance Local anesthetic mixture will be administered by multi injection method between the nerve groups seen in the sonoanatomical image.
  Arms: multi
Procedure: diagraphma muscle evaluation with ultrasound — All patients will be evaluated with USG in a head-up position facing the side to be operated before and 30 minutes after the block is performed.
  The probe will be placed perpendicular to the chest wall, in the eighth or ninth intercostal space, between the anterior axillary and midaxillary lines, 0.5 to 2 cm below the costophrenic sinus.

SUMMARY:
Brachial plexus blocks used for anesthesia in upper extremity operations can be performed with interscalene, axillary, supraclavicular and infraclavicular approaches.

Plexus blockage can be performed under the guidance of needle nerve stimulation, artery palpation or ultrasonography (USG).

Nowadays, the simultaneous use of USG during the block allows the protection of structures such as nerves, pleura and vessels, and allows practitioners to see the needle and the spread of local anesthetic during the injection.

Although supraclavicular block seems to be advantageous because the brachial plexus is more compact and superficial in this region, it has a disadvantage of being close to the pleura. (Increased risk of pneumothorax) With the use of USG, this risk has decreased and the supraclavicular block has become an alternative to infraclavicular block, which is widely used in upper extremity surgery.

Due to the compact structure of the brachial plexus trunk at the first rib level, the application of the block is easier and the block formation is faster due to the peripheral spread of the local anesthetic.

With the spread of local anesthetic to C3-C5 nerve roots in the brachial plexus, paralysis can be seen in the ipsilateral phrenic nerve up to 67%. Patients who will be operated on, especially in patients with respiratory distress, may experience respiratory distress due to the dysfunction of that side diaphragm muscle. With the help of ultrasound, the inspiratory and end-expiratory thickness of the diaphragm is measured with the Diaphragm Thickness Index (DTI), which is a new and effective method used as a mechanical ventilator weaning index in intensive care units. With this method, we can examine the effect of phrenic nerve block on diaphragm muscle due to local anesthesia in the acute period.

DTI is calculated as a percentage from the following formula:

(Max thickness at the end of inspiration - Max thickness at the end of the expiration) / Max thickness at the end of the expiration. By comparing 3 different approaches used in supraclavicular block, we aimed to investigate the most appropriate block approach in terms of effectiveness, speed, complication rate, effects on diaphragm and 6 months effects.

DETAILED DESCRIPTION:
In this prospective randomized double-blind study, patients will be divided into 3 groups using a computer program.

Standard monitoring (ECG, pulse oximetry, noninvasive blood pressure) will be applied to the patients who will then be taken to the block application room . After the peripheral vascular access is established on the hand that will not be operated on, premedication will be provided with 2 mg iv midazolam.

The blocks will be performed by an experienced anesthesiologist with the USG guidance. Block evaluation and measurements will be made by a different experienced anesthesiologist. After the antisepsis of the area to be blocked, a 22G 50 mm stimulator needle will be used for the block. Intermittent negative aspiration will be performed during all procedures to detect possible vascular puncture. The local anesthetic mixture we routinely use in our clinic will be used. 20 ml of bupivacaine(Buvicaine HCl %0.5) and prilocaine(Priloc HCl %2) 1:1 mixture will be prepared in a way that there will be 5mcg adrenaline per ml.(9ml bupivacaine, 9ml prilocaine and 2ml saline with 50 mcg adrenaline per ml) The ultrasound probe will be placed on the clavicle, the supraclavicular block will be applied in the coronal oblique plane using the in-plane technique.

3 different approaches of supraclavicular block will be compared. Approaches share the same probe position and needle entry point but differ in where the local anesthetic is given.

Group 1: Local anesthetic mixture will be given to the corner pocket - where the artery and the first rib intersect in the sonoanatomical image.

Group 2: 10 ml of the local anesthetic mixture will be given to the described corner pack and the remaining 10 ml into the largest nerve cluster (Intracluster injection).

Group 3: Local anesthetic mixture will be administered by multi injection method between the nerve groups seen in the sonoanatomical image.

The diaphragm thickening fraction and evaluations will be made by another experienced anesthesiologist, double-blindness will be achieved by being blind to the patient's group.

Effects of phrenic nerve block on diaphraghma muscle will be evaluated by diaphraghma thickining fraction.All patients will be evaluated with USG in a head-up position facing the side to be operated before and 30 minutes after the block is performed.The probe will be placed perpendicular to the chest wall, in the eighth or ninth intercostal space, between the anterior axillary and midaxillary lines, 0.5 to 2 cm below the costophrenic sinus.

The diaphragm will be viewed as a structure with three distinct layers, including two parallel echoic lines (Diaphragmatic pleura and peritoneum) and a hypoechoic line between them (Diaphragm muscle) . The patient will be instructed to breathe up to total lung capacity (TLC) and then exhale to residual volume (RV).

Several diaphragm images will be taken, at least three at the point of maximum thickening in TLC and at least three at minimum thickness in RV.

On each B-mode image, diaphragm thickness will be measured from the middle of the pleural line to the middle of the peritoneal line. Then DTI will be calculated as a percentage from the following formula:

(Max thickness at the end of inspiration - Max thickness at the end of the expiration) / Max thickness at the end of the expiration.

With this formula, we can determine the involvement of phrenic nerve by looking at the rate of diaphragm thickening before and after supraclavicular block in different groups.

As a first line rescue anesthesia, patients will receive sedoanalgesia with remifentanil infusion. Laryngeal mask and general anesthesia will be commenced if needed. The postoperative analgesic regimen will routinely contain 1000 mg IV acetaminophen (3x1) and, if necessary, 1 mg opioid (Tramadol) per kg will be given.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled scheduled for hand, wrist, forearm, arm surgery
* Patients who has informed consent for study
* Patients with American Society of Anesthesiologists Physical Status Classification(ASA) I,II and III

Exclusion Criteria:

* Patient's refusal to participate
* Patients under 18 years of age
* Patients with known local anesthetic allergy
* Patients with Body mass index> 35
* Patients diagnosed sepsis and bacteriemia,
* Skin infection at the injection site,
* History of coagulopathy or anticoagulant therapy
* Patients with uncontrolled diabetes,
* Uncoordinated patients,
* Psychological and emotional lability,
* Patients with anatomical disorders at application points
* Pregnant patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Comparison of Three Different Approach for Supraclavicular Blocks Effects on Diaphragm Thickening Fraction | Comparison of Diaphragm Thickening Fraction will be evaluated 30 minutes after the block is performed.
  Several diaphragm images will be taken, at least three at the point of maximum thickening in TLC and at least three at minimum thickness in RV. On each B-mode image, diaphragm thickness will be measured from the middle of the pleural line to the middle of the peritoneal line. Then DTI will be calculated as a percentage from the formula: (Max thickness at the end of inspiration - Max thickness at the end of the expiration) / Max thickness at the end of the expiration. All patients will be evaluated with USG in a head-up position facing the side to be operated 30 minutes after the block is performed.

SECONDARY OUTCOMES:
The sensory block level | Following the block operation, the sensory block level will be recorded at the 5th, 10th, 15th, 20th, 25th and 30th minutes
  Sensory block level; The level of block that will occur in the sensory areas of axillary, median, radial, ulnar, musculocutaneous, cutaneous brachia and cutaneous antebraki medialis nerves will be evaluated by performing a pinprick test and its level will be recorded (0 = Painful, no block; 1 = Partial block-analgesia, only feeling of touch; 2 = Complete block, no pain).
The motor block level | Following the block operation, the motor block level will be recorded at the 5th, 10th, 15th, 20th, 25th and 30th minutes
  It will be evaluated with the Modified Bromage scale:
  0 = No blocks, he can lift his arm,
  1= Motor power is low but the arm is movable, 2 = The arm is immobile but the fingers are movable, 3 = Complete block, no movement in hand or arm
Block success | At the 30th minute of LA application,
  It will be defined as the presence of the pinprick test in the musculacutaneous, radial, ulnar, median, cutaneous antebraki nerves with no pain or only feeling of touch. If any of these nerves are not blocked, it will be considered a failed block.
Postoperative analgesia time | The hour when NRS> 1 in the first 24 hours will be recorded.
  Numeric rating scale; patient values pain between 0 and 10; 0 = No pain-10 = Intractable pain
Pain Score Follow-up | 2nd, 6th, 12th and 24th hours
  Numeric rating scale; patient values pain between 0 and 10; 0 = No pain-10 = Intractable pain
Block return time | The return time of sensory and motor block will be recorded within the first 24 hours.
  Sensory (the time from local anesthetic injection until the patient fully perceives the upper limb) and motor (the time from local anesthetic injection to the moment the patient's upper limb regains muscle strength) will be recorded as the time to return the block.
Block application time | intraoperative (during block application)
  It will be defined as the time from the moment the needle passes through the skin until the local anesthetic is given and the needle is withdraw.
Block onset time | baseline (before surgery)
  It will be defined as the time required to initiate anesthesia and analgesia in all 5 distal nerves from the local anesthetic injection.
Patient and surgeon satisfaction | immediately after the surgery
  Patient and surgeon satisfaction will be evaluated as: 1 = Complete dissatisfaction, 2 = Moderate satisfaction, 3 = Full satisfaction after the procedure.
Undesirable side effects: | Patients will be observed for 24 hours,
  Recorded when there is vascular puncture, hematoma, signs of LA toxicity, respiratory distress, pneumothorax, and Horner Syndrome.
The first opioid requirement hour | If pain occurs within the first 24 hours from the time the block transaction ends.
  The first hour of opioid requirement of the patients will be recorded.(When NRS> 3) Opioids(Tramadol) will be administered to patients in case demanded.
24-hour total opioid consumption | It will be defined as 24 hours from the time the block transaction ends.
  It will be recorded how much opioid he needs to use for 24 hours.Opioids(Tramadol) will be administered to patients in case demanded.
Chronic pain questionnaire | 6 months after operation
  After 6 months, patients will be called and questioned by phone.

CONTACTS AND LOCATIONS:
Overall Officials: Çağrı Yeşilnacar, MD, Study Chair — Izmir Bozyaka Training and Research Hospital; Zeki T Tekgül, Assoc Prof, Study Chair — Izmir Bozyaka Training and Research Hospital; AYSUN A KAR, MD, Study Chair — Izmir Bozyaka Training and Research Hospital; TAŞKIN ALTAY, Assoc Prof, Study Chair — Izmir Bozyaka Training and Research Hospital
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Izmir, Karabaglar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrari G, De Filippi G, Elia F, Panero F, Volpicelli G, Apra F. Diaphragm ultrasound as a new index of discontinuation from mechanical ventilation. Crit Ultrasound J. 2014 Jun 7;6(1):8. doi: 10.1186/2036-7902-6-8. eCollection 2014. PMID 24949192
- [Background] Petrar SD, Seltenrich ME, Head SJ, Schwarz SK. Hemidiaphragmatic paralysis following ultrasound-guided supraclavicular versus infraclavicular brachial plexus blockade: a randomized clinical trial. Reg Anesth Pain Med. 2015 Mar-Apr;40(2):133-8. doi: 10.1097/AAP.0000000000000215. PMID 25650633
- [Background] Renes SH, Spoormans HH, Gielen MJ, Rettig HC, van Geffen GJ. Hemidiaphragmatic paresis can be avoided in ultrasound-guided supraclavicular brachial plexus block. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):595-9. doi: 10.1097/aap.0b013e3181bfbd83. PMID 19916254